CLINICAL TRIAL: NCT04476875
Title: Patient-controlled Outpatient Follow-up on Demand for Patients With Rheumatoid Arthritis: a Two-year Randomized Trial
Brief Title: Outpatient Follow-up on Demand in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, René Panduro Poggenborg, Principal Investigator, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Protokol-38787-v1-08072013
Record Dates: First submitted 2020-07-07; First posted 2020-07-20 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Follow-up on demand
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Observation of clinical outcomes in two groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open outpatient clinic programme (OOCP) (Active Comparator): OOCP patients had no scheduled appointments but were allowed acute appointments with their rheumatologist, and had access to nurse-led consultations and telephone helpline.
  Interventions: Other: Open Outpatient Clinic Programme
- Traditional scheduled routine follow up (TSRF) (No Intervention): Appointments for the TSRF group were scheduled according to routine procedures.

INTERVENTIONS:
Other: Open Outpatient Clinic Programme
  Arms: Open outpatient clinic programme (OOCP)

SUMMARY:
A two-year randomized controlled trial with rheumatoid arthritis (RA) patients. Patients were randomized electronically with stratification according to biologic and non-biologic treatment to the open outpatient clinic programme, or usual care. Patients were evaluated at baseline, year 1 and 2, including assessment of disease activity and reporting of outcomes measures on a touch screen at the clinic.

DETAILED DESCRIPTION:
A two-year randomized controlled trial with rheumatoid arthritis (RA) patients. At baseline, patients were randomized electronically with stratification according to biologic and non-biologic treatment to the open outpatient clinic programme, or usual care. Patients were evaluated at baseline, year 1 and 2, including assessment of disease activity (DAS-28), blood tests, bone erosions on plain radiographs of hands and feet, and patient reported outcome measures.

The objective of the study was to compare an outpatient system for Danish RA patients based on patient self-controlled outpatient follow up on demand, Open Outpatient Clinic Programme with traditional scheduled routine follow-up regarding patient satisfaction and effect on traditional disease markers.

The Danish National Patient Registry (DANBIO) was used to identify eligible patients with RA. At pre-planned routine visits with the rheumatologist, identified patients were screened according to inclusion and exclusion criteria.

The intervention group had no scheduled appointments at the outpatient clinic, but they could book acute appointments with their contact rheumatologist within 5 days or less whenever they deemed it necessary. They also had access to nurse-led consultations without pre-booked appointments and to a nurse-led telephone helpline

ELIGIBILITY:
Inclusion Criteria:

RA. Disease duration of at least 1 year.

Exclusion Criteria:

Patients treated with monthly intravenous biological medicine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue Scale (VAS) Patient satisfaction | 2 years
  Patient reported outcome which assess overall how satisfied the patient is regarding the management of their rheumatoid arthritis in the hospital setting. Patient satisfaction is scored on a visual analogue scale (VAS). Minimum score is 0 (worst), and maximum score 100 (best).

SECONDARY OUTCOMES:
Disease activity score in 28 joints (DAS28) | 2 years
  DAS28 is a measure of disease activity in rheumatoid arthritis. To calculate the DAS28 we counted the number of swollen joints and tender joints (out of the 28), measured C reactive protein (CRP) and assessed the patients 'global assessment of health' (indicated on a visual analogue scale from 0 (best) to 100 (worst)
Radiographic progression | 2 year
  Radiographs of hands and feet were compared between baseline and follow-up, regarding development of structural changes, including bone erosions. A musculoskeletal radiologist evaluated whether erosive development or progression was present.

CONTACTS AND LOCATIONS:
Overall Officials: Annette Hansen, Study Chair — University Hospital Gentofte
Locations (1):
- University Hospital Gentofte, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poggenborg RP, Madsen OR, Sweeney AT, Dreyer L, Bukh G, Hansen A. Patient-controlled outpatient follow-up on demand for patients with rheumatoid arthritis: a 2-year randomized controlled trial. Clin Rheumatol. 2021 Sep;40(9):3599-3604. doi: 10.1007/s10067-021-05674-y. Epub 2021 Mar 6. PMID 33677724